CLINICAL TRIAL: NCT04314115
Title: Prevention of Mental Health Problems in People Exposed to a Recent Highly Stressful Event: a Randomized Controlled Study
Brief Title: Prevention of Mental Health Problems in People Exposed to a Recent Highly Stressful Event.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas, Chile (Other)
Collaborators: Universidad de Concepcion (Other)
Responsible Party: Principal Investigator, Felipe E. García, Principal investigator, Universidad Santo Tomas, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1180134
Record Dates: First submitted 2020-03-09; First posted 2020-03-19 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Posttraumatic Stress Disorder; Acute Post-Traumatic Stress Disorder; Depressive Symptoms
Keywords: Mindfulness; Brief systemic therapy; Cognitive Behavioral Therapy; Mental health; Prevention; Stressful events; Post-traumatic symptoms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Psychological Well-Being | interventions — Mindfulness; Crisis Intervention; Methods; Cognitive Behavioral Therapy; Psychology, Positive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness (Active Comparator): A brief intervention in mindfulness will be administered
  Interventions: Other: Mindfulness
- Systemic therapy (Active Comparator): A brief systemic therapy intervention will be administered
  Interventions: Other: Systemic therapy
- Cognitive behavioral therapy and positive psychology (Active Comparator): A brief intervention of traditional cognitive behavioral therapy with positive psychology elements will be administered
  Interventions: Other: Cognitive behavioral therapy and positive psychology
- Waiting list (No Intervention): Waiting list, as a control group

INTERVENTIONS:
Other: Mindfulness — Brief intervention in mindfulness, of individual type, of four sessions of sixty minutes per week, in addition to individual tasks, according to protocol of brief intervention in developed mindfulness.
  Other Names: Brief intervention in mindfulness
  Arms: Mindfulness
Other: Systemic therapy — Brief systemic therapy intervention, of four weekly sessions of sixty minutes, with individual tasks and assignments, according to the protocol designed.
  Other Names: Intervention in brief systemic therapy
  Arms: Systemic therapy
Other: Cognitive behavioral therapy and positive psychology — Brief intervention of traditional cognitive behavioral therapy with elements of positive psychology, of four weekly sessions of sixty minutes, with individual assignments and assignments, according to the protocol designed.
  Other Names: Brief intervention of traditional cognitive behavioral therapy and positive psychology
  Arms: Cognitive behavioral therapy and positive psychology

SUMMARY:
This project evaluates the effectiveness of three intervention models for the prevention of mental health problems in people who have suffered a recent highly stressful event, through an experimental design, with a control group and random assignment of participants in each group .

The preventive interventions that will be evaluated will be based on three different psychotherapeutic models: brief systemic therapy, cognitive behavioral therapy and mindfulness.

It is expected to observe a significant reduction in post-traumatic and depressive symptoms, and an increase in subjective well-being and post-traumatic growth, compared to the control group. In addition, the moderating effect of psychological processes such as cognitive rumination, emotional self-regulation and coping strategies used in the relationship between the type of intervention and its results will be evaluated.

If the hypotheses are confirmed, this study will allow the prevention of emotional distress associated with a highly stressful event, as well as the promotion of positive results, through empirically supported, low-cost strategies and with results that are capable of demonstrating their effectiveness.

DETAILED DESCRIPTION:
Highly stressful events are alterations in the life history of an individual that require an adaptation effort. Available studies warn that about 82 to 90% of the general population will be exposed to some type of traumatic event at some time in their lives. Chile, for example, is constantly prone to suffer highly stressful events of massive order, due to the high frequency of natural disasters that affect it from time to time: earthquakes, volcanic eruptions, floods, floods, as well as stressors that individually affect such as criminal violence, sexual abuse or threatening diseases. This makes the probability that a person has to be exposed to an event of this type is high, developing from it various consequences.

Although the majority will not develop long-term negative consequences, a significant percentage may develop different mental health problems, such as post-traumatic symptoms, and depression. It is estimated, for example, that 25% of people exposed to the 2010 Chile earthquake in the Bío Bío region developed a post-traumatic stress disorder. Likewise, 13.5% of adolescents exposed to the same earthquake developed high levels of depressive symptomatology.

However, there are also more adaptive responses after living these events, one of them is to grow from the negative experience. This possibility has been called posttraumatic growth [PTG], defined as the perception of positive changes that a person experiences as a result of the process of fighting a trauma. Although this growth is the result of an event that caused people to feel unwell, which explains the high relationship between PTSD and PTG in some cross-sectional studies, in multivariate studies and longitudinal different predictors are observed, and in prospective studies it has been determined that the highest PTG is associated in the long term with a higher level of well-being and a decrease in posttraumatic and depressive symptomatology, as well as a better quality of life.

Prevention and promotion actions are gaining increasing importance in all areas of the health field, including difficulties that occur in emergencies and post-emergencies. It is therefore important to determine the factors that contribute to a higher level of subjective well-being and PTG or a lower level of post-traumatic or depressive symptoms after experiencing a highly stressful event. Research that has been conducted to determine the predictors of these responses has shown their association with perceived severity, rumination, emotional self-regulation, religious coping or other coping strategies, such as the search for social support and the active coping.

In a study carried out by García in 2016-2017 with people facing a highly stressful event such as an accident at work intrusive rumination, brooding, deliberate rumination were determined as early predictors of posttraumatic symptomatology. Subjective severity of the event, negative religious coping and positive reinterpretation (inverse predictor), brooding, negative religious coping and positive religious coping (reverse predictor) were determined as early predictors of depressive symptomatology. Regarding positive responses, deliberate rumination and positive religious coping were determined as predictors of PTG, but only initial well-being was a predictor of subsequent subjective well-being. The strength of this study is that it evaluated the predictors less than a month after the event occurred, and continued its evolution at six months and one year after the accident occurred. Thus arises the possibility, supported by current empirical data, to develop intervention programs that encourage cognitive reassessment, deliberate rumination on the event, positive religious coping, active coping, the search for social support and initial well-being, in addition to reduce expressive suppression, intrusive and negative rumination, and negative religious confrontation.

Prevention is one of the most effective ways to reduce the prevalence of mental health problems, as it aims to reduce risk factors, strengthen protective factors and reduce psychiatric symptoms and disability, as well as early onset of some symptoms of mental disorders; It also improves positive mental health, contributes to better physical health and generates social and economic benefits. The prevention of mental disorders focuses on those determinants that exert a causal influence. Those preventive interventions aimed at strengthening protection factors often overlap with mental health promotion.

Regarding the prevention of post-traumatic symptoms, available studies show interventions aimed at earthquake survivors, serious or terminal diseases, wars and violations, among others.

From a cognitive-behavioral approach, techniques have been proposed aimed at increasing coping resources both instrumental and emotional as well as self-regulation capacity and relaxation training.

In a recent study with a non-clinical population, Mindfulness was used in a four-session intervention, with a decrease in depressive symptomatology, an increase in subjective well-being, as well as a reduction in emotional suppression and rumination and an increase in Cognitive reevaluation as an emotional regulation strategy. The size of the intervention effect was a d-Cohen of 0.65 for depressive symptomatology and 0.64 for psychological well-being, both of average value.

Regarding the brief systemic approach, strategies aimed at strengthening personal resources, resignifying negative experiences, reconnecting with social networks, as well as facilitating emotional expression have been proposed. These strategies were used in women newly diagnosed with breast cancer, through a four-session workshop, obtaining a reduction at the end of the post-traumatic symptomatology intervention, depressive symptomatology and physical discomfort associated with the disease. In this study, the effect size was a d-Cohen of 1.30 for post-traumatic symptomatology and 0.57 for depressive symptomatology, considered high and medium values, respectively.

Given the background presented, it is crucial to develop research that can shed light on the challenges related to the prevention of emotional distress associated with a highly stressful event, such as those that frequently affect the Chilean population, as well as with the promotion of positive results, through empirically backed strategies, of low cost and with results that are capable of demonstrating their effectiveness.

Such interventions will allow early response programs to be implemented in case of massive events, such as natural disasters.

HYPOTHESIS

1. Brief preventive interventions reduce levels of post-traumatic symptoms, and also reduce depressive symptoms and increase levels of post-traumatic growth and subjective well-being in people recently exposed to a highly stressful event.
2. The available preventive models (cognitive-behavioral, mindfulness and brief systemic) have similar and superior results to the control group (waiting list) for the reduction of post-traumatic symptomatology, in addition to the reduction of depressive symptomatology and the increase of growth levels and subjective well-being in people recently exposed to a highly stressful event.
3. The changes produced in the levels of posttraumatic and depressive symptomatology, posttraumatic growth and subjective well-being are maintained six months after the intervention.
4. Changes in the levels of subjective severity of the event, mental rumination, coping strategies and emotional self-regulation mediate the outcome of the interventions.

OVERALL OBJECTIVE Evaluate three brief intervention programs in individual format (cognitive-behavioral, mindfulness and brief systemic) for the prevention of post-traumatic and depressive symptomatology and the promotion of subjective well-being and post-traumatic growth in people who have been exposed to a recent highly stressful event.

SPECIFIC OBJECTIVES

1. Evaluate the effect of brief preventive interventions on posttraumatic symptomatology in people who have been exposed to a recent highly stressful event, at the end of treatment and six months after the intervention.
2. Evaluate the effect of brief preventive interventions on depressive symptomatology, posttraumatic growth and subjective well-being, at the end of treatment and at six months.
3. Evaluate the mediation of changes in cognitive rumination, coping strategies and emotional self-regulation between the intervention and its effect on post-traumatic and depressive symptomatology, post-traumatic growth and subjective well-being.

DESIGN A randomized experimental design of parallel groups will be used, with three randomized intervention modalities and a control group, with repeated measures through pre and post intervention evaluation and follow-up at six months.

PROCESS

The procedure will be divided into three main phases:

A) development of intervention protocols, B) evaluation of the protocols in pilot intervention, C) randomized clinical trial.

A) Development of intervention protocols. For this phase, an exhaustive review of the research literature will be carried out first to examine preventive interventions that have pointed to the decrease in post-traumatic or depressive symptoms or to the promotion of subjective well-being or PTG in the population that has been exposed to a highly stressful or potentially traumatic events. From this review of the literature, interventions will be extracted to be included in individual treatment programs of four sessions for each modality, which will be organized in a treatment manual.

B) Evaluation of the protocols in pilot intervention. Individual intervention pilots will be executed with a small number of participants, 12 in total, 4 for each program, one program for each region in which it will be implemented (Antofagasta, Maule and Bío-Bío). To do this, the following steps will be used: a) selection of therapists, who must demonstrate prior training at the level of courses, graduates or any certified instance in any of the three intervention models to be used, b) training of therapists in the protocol of intervention, both theoretical and expository, as well as through guided exercises, role play and video analysis of their own interventions, c) selection of participants according to the inclusion and exclusion criteria defined, d) pre-intervention evaluation, the defined instrument battery being applied to the participants, e) application of the intervention for four sessions, which will be videotaped, g) application of the post-intervention instrument battery, g ) semi-structured interviews with therapists, to establish adjustments to the program used considering their experience in the application of the same, h) analysis of the videos of the interventions, and i) elaboration of the definitive protocols.

C) Randomized clinical trial Prior to the clinical trial, a dissemination campaign will be carried out in the universities of each city, in order to increase the number of people susceptible to receiving care. For the intervention itself, the CONSORT protocol will be followed for randomized clinical trials. The final intervention protocols will be executed for 160 participants, 40 for each intervention program and 40 for the control group on the waiting list. To do this, the following steps will be used: a) inclusion of therapists who participated in the pilot trial, and training of new therapists, who meet the requirements outlined in the previous section, in the intervention protocols, b) evaluation of depressive symptomatology and post-traumatic, because given the preventive nature of the interventions, people with high levels in these cadres will not participate in the study and will be referred to free psychological care in the sponsoring universities, c) randomization to the 3 types of intervention and control group, using ad-hoc software, d) pre-intervention evaluation, e) application of the intervention, 25% of which will be videotaped, in order to ensure the fidelity of the intervention and supervise the Therapists, f) post-intervention evaluation, g) follow-up (at six months). In the case of the control group on the waiting list, they will start the intervention four weeks after their first evaluation, in order to have a comparison group without intervention in the second measurement. However, when intervened after the fourth week (once again randomizing the type of intervention), there will be no control group for follow-up. This for ethical reasons, because you cannot leave someone who requires it without the support that the rest of the participants receive. In addition, those who show high rates of discomfort at follow-up will also be referred to free psychotherapy in the sponsoring universities.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be to be of legal age and to have lived the highly stressful experience in the last three months (a check-list of events will be available).

Exclusion Criteria:

* Those who have already been previously given psychological care will be excluded due to the consequences generated by the same event and who, due to their health condition, are prevented from receiving individual care in the first three months after the event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Post-traumatic symptoms, pre-intervention evaluation | Pre-intervention evaluation
  It will be measured with the brief post-traumatic stress disorder qualification interview (SPRINT-E scale) (Norris, Hamblen, Brown & Schinka, 2008), validated for the Chilean population by Leiva and Gallardo (2013), which has 14 items. Its minimum score is 0 and its maximum score is 36. A higher score means that the patient is worse, due to high post-traumatic symptoms.
Post-traumatic symptoms, post intervention evaluation | Post-intervention evaluation, four weeks after the start of the intervention.
  It will be measured with the brief post-traumatic stress disorder qualification interview (SPRINT-E scale) (Norris, Hamblen, Brown & Schinka, 2008), validated for the Chilean population by Leiva and Gallardo (2013), which has 14 items. Its minimum score is 0 and its maximum score is 36. A higher score means that the patient is worse, due to high post-traumatic symptoms.
Post-traumatic symptoms, follow-up measure | Follow-up measurement six months after the end of the intervention.
  It will be measured with the brief post-traumatic stress disorder qualification interview (SPRINT-E scale) (Norris, Hamblen, Brown & Schinka, 2008), validated for the Chilean population by Leiva and Gallardo (2013), which has 14 items. Its minimum score is 0 and its maximum score is 36. A higher score means that the patient is worse, due to high post-traumatic symptoms.

SECONDARY OUTCOMES:
Depressive symptomatology | A pre-intervention evaluation will be performed before starting the intervention, a post-intervention measurement four weeks later, and a follow-up measurement six months after the end of the intervention.
  To measure depressive symptoms, the Depression Scale of the Center for Epidemiological Studies will be used: Center for Epidemiological Studies - depression (CES-D; Radloff, 1977, translated by Gempp, Avendaño and Muñoz, 2004), which has 20 items. The lowest score is 0 and the highest is 60. A lower score means an improvement due to the fact that the patient has decreased depressive symptoms, while a higher score means that the patient feels worse due to the greater depressive symptoms.
Posttraumatic growth | A pre-intervention evaluation will be performed before starting the intervention, a post-intervention measurement four weeks later, and a follow-up measurement six months after the end of the intervention.
  To measure post-traumatic growth, the Post-traumatic Growth Inventory - Short Format Scale (PTGI-SF; Tedeschi and Calhoun, 1996), validated for Chile by García and Wlodarczyk (2015), which has 10 items, will be used. The lowest score is 0 and the highest is 50. A higher score means that the patient has experienced improvement due to increased post-traumatic growth.
Subjective well-being | A pre-intervention evaluation will be performed before starting the intervention, a post-intervention measurement four weeks later, and a follow-up measurement six months after the end of the intervention.
  It will be measured with the Life Satisfaction Scale (Diener, Emmos and Griffin, 1985), validated in Spanish by Moyano and Ramos (2007), which has 5 items. The lowest score is 5 and the highest is 35. A higher score means an improvement in the patient due to greater satisfaction with life.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Santo Tomas, Concepción, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez AR, Estario JC, Enders JE, Neira MJ, Abeldano RA. [Screening for posttraumatic stress disorder in people affected by the 2010 earthquake in Chile.]. Cad Saude Publica. 2014 Nov;30(11):2377-2386. doi: 10.1590/0102-311x00141313. Spanish. PMID 25493991
- [Background] Alarcón, R. (2002). Trastorno por estrés postraumático: estudios en veteranos de guerra norteamericanos y su relevancia para América Latina. Revista Chilena de Neuro-psiquiatría, 40, 35-47.
- [Background] Altindag A, Ozen S, Sir A. One-year follow-up study of posttraumatic stress disorder among earthquake survivors in Turkey. Compr Psychiatry. 2005 Sep-Oct;46(5):328-33. doi: 10.1016/j.comppsych.2005.01.005. PMID 16122532
- [Background] Alzugaray, C., García, F., Reyes, A., & Álvarez, R. (2015). Propiedades psicométricas de una versión breve de la escala de rumiación relacionada a un evento en población chilena afectada por eventos altamente estresantes. Ajayu, 13(2), 183-198.
- [Background] Amutio-Kareaga A, Garcia-Campayo J, Delgado LC, Hermosilla D, Martinez-Taboada C. Improving Communication between Physicians and Their Patients through Mindfulness and Compassion-Based Strategies: A Narrative Review. J Clin Med. 2017 Mar 17;6(3):33. doi: 10.3390/jcm6030033. PMID 28304333
- [Background] Andrades, M., García, F., Calonge. I., & Martínez-Arias, R. (2017). Posttraumatic growth in children and adolescents exposed to the 2010 earthquake in Chile and its relationship with rumination and posttraumatic stress symptoms. Journal of Happiness Studies, 1-13.
- [Background] Andrades M, Garcia FE, Reyes-Reyes A, Martinez-Arias R, Calonge I. Psychometric properties of the Posttraumatic Growth Inventory for Children in Chilean population affected by the earthquake of 2010. Am J Orthopsychiatry. 2016;86(6):686-692. doi: 10.1037/ort0000182. Epub 2016 May 23. PMID 27213218
- [Background] Avilés, P., Cova, F., Bustos, C., & García, F.E. (2014). Afrontamiento y rumiación frente a eventos adversos y crecimiento postraumático en estudiantes universitarios. Liberabit, 20(2), 281-292.
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Basoglu M, Livanou M, Salcioglu E. A single session with an earthquake simulator for traumatic stress in earthquake survivors. Am J Psychiatry. 2003 Apr;160(4):788-90. doi: 10.1176/ajp.160.4.788. PMID 12668372
- [Background] Beyebach, M. (2006). 24 ideas para una psicoterapia breve. Barcelona: Herder.
- [Background] Beyebach, M. (2014). Change factors in solution-focused brief therapy: A review of the Salamanca studies. Journal of Systemic Therapies, 33(1), 62-77.
- [Background] Breslau N. Epidemiologic studies of trauma, posttraumatic stress disorder, and other psychiatric disorders. Can J Psychiatry. 2002 Dec;47(10):923-9. doi: 10.1177/070674370204701003. PMID 12553127
- [Background] Breslau N, Kessler RC, Chilcoat HD, Schultz LR, Davis GC, Andreski P. Trauma and posttraumatic stress disorder in the community: the 1996 Detroit Area Survey of Trauma. Arch Gen Psychiatry. 1998 Jul;55(7):626-32. doi: 10.1001/archpsyc.55.7.626. PMID 9672053
- [Background] Cann A, Calhoun LG, Tedeschi RG, Triplett KN, Vishnevsky T, Lindstrom CM. Assessing posttraumatic cognitive processes: the Event Related Rumination Inventory. Anxiety Stress Coping. 2011 Mar;24(2):137-56. doi: 10.1080/10615806.2010.529901. PMID 21082446
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Chaves, C., Hervás, G. & García, F. & Vázquez, C. (2015). Building life satisfaction through well-being dimensions: A longitudinal study in children with a life-threatening illness. Journal of Happiness Studies, 17(3), 1051-1067.
- [Background] Cova, F., Rincón, P., & Melipillán, R. (2009). Reflexión, rumiación negativa y desarrollo de sintomatología depresiva en adolescentes de sexo femenino. Terapia Psicológica, 27(2), 155-160.
- [Background] Gómez, A. & Cárdenas, G. (2016). Reacciones postraumáticas: revisión desde una perspectiva dimensional. Psicología Iberoamericana, 24(1), 70-79.
- [Background] Creamer M, McFarlane AC, Burgess P. Psychopathology following trauma: the role of subjective experience. J Affect Disord. 2005 Jun;86(2-3):175-82. doi: 10.1016/j.jad.2005.01.015. PMID 15935237
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Díaz, C. A., Quintana, G. R., & Vogel, E. H. (2012). Síntomas de depresión, ansiedad y estrés posttraumático en adolescentes siete meses después del terremoto del 27 de febrero de 2010 en Chile. Terapia Psicológica, 30(1), 37-43.
- [Background] García, F. (2013). Terapia sistémica breve. Fundamentos y aplicaciones (1ra. edición). Santiago de Chile: RIL.
- [Background] García, F. & Ceberio, M.R. (2016). Manual de terapia sistémica breve. Santiago de Chile: Mediterráneo.
- [Background] García, F., Cova, F. & Melipillán, R. (2013). Propiedades psicométricas del Inventario de Crecimiento Postraumático en población chilena afectada por un desastre natural. Revista Mexicana de Psicología, 30 (2), 145-153.
- [Background] Garcia FE, Cova F, Rincon P, Vazquez C. Trauma or growth after a natural disaster? The mediating role of rumination processes. Eur J Psychotraumatol. 2015 Jul 31;6:26557. doi: 10.3402/ejpt.v6.26557. eCollection 2015. PMID 26234365
- [Background] Garcia FE, Duque A, Cova F. The four faces of rumination to stressful events: A psychometric analysis. Psychol Trauma. 2017 Nov;9(6):758-765. doi: 10.1037/tra0000289. Epub 2017 Jun 8. PMID 28594202
- [Background] García, F. & Ilabaca, D. (2013). Ruptura de la pareja, afrontamiento y bienestar psicológico en adultos jóvenes. Ajayu, 11(2), 157-172.
- [Background] García, F., Jaramillo, C., Martínez, A.M., Valenzuela, I. & Cova, F. (2014). Respuestas psicológicas ante un desastre natural: Estrés y crecimiento postraumático. Liberabit, 20, 121-130.
- [Background] García, F. & Mardones, R. (2010). Prevención de trastorno de estrés postraumático en supervivientes del terremoto de Chile de febrero de 2010: una propuesta de intervención narrativa. Terapia psicológica, 28(1), 85-93.
- [Background] García, F., Páez, D., Cartes, G., Neira, H. & Reyes, A. (2014). Religious coping, social support and subjective severity as predictors of posttraumatic growth in people affected by the earthquake in Chile on 27/F 2010. Religions, 5, 1132-1145.
- [Background] García, F., Páez, D., Reyes, A. & Álvarez, R. (2017). Religious coping as moderator of psychological responses to stressful events: A longitudinal study. Religions, 8(62), 1-13.
- [Background] García, F. & Rincón, P. (2011). Prevención de sintomatología postraumática en mujeres diagnosticada con cáncer de mama: Evaluación preliminar de un modelo de intervención narrativo. Terapia Psicológica, 29(2), 175-183.
- [Background] García, F. & Wlodarczyk, A. (2015). Psychometric Properties of the Post-traumatic Growth Inventory - Short Form among Chilean Adults. Journal of Loss and Trauma. 21(4), 303-314.
- [Background] García, F., Wlodarczyk, A., Reyes, A., San Cristóbal, C. & Solar, C. (2014). Violencia en la pareja, apoyo social y bienestar psicológico en adultos jóvenes. Ajayu, 12 (2), 246-265.
- [Background] García-Campayo, J. & Demarzo, M. (2015). Mindfulness y compasión: La nueva revolución. Barcelona: Siglantama.
- [Background] Gempp, R., Avendaño, C., & Muñoz, C. (2004). Normas y punto de corte para la Escala de Depresión del Centro para Estudios Epidemiológicos (CES-D) en población juvenil chilena. Terapia Psicológica, 22(2), 145-156.
- [Background] Gross JJ, John OP. Individual differences in two emotion regulation processes: implications for affect, relationships, and well-being. J Pers Soc Psychol. 2003 Aug;85(2):348-62. doi: 10.1037/0022-3514.85.2.348. PMID 12916575
- [Background] Guerra, C., & Plaza, H. (2009). Tratamiento Cognitivo-Conductual del Estrés Postraumático en un caso de violación infantil. Revista de Psicología, 18(1), 103-129.
- [Background] Kuoppala J, Lamminpaa A, Vaananen-Tomppo I, Hinkka K. Employee well-being and sick leave, occupational accident, and disability pension: a cohort study of civil servants. J Occup Environ Med. 2011 Jun;53(6):633-40. doi: 10.1097/JOM.0b013e31821aa48c. PMID 21654433
- [Background] Leiva-Bianchi, M.C., & Gallardo, I. (2013). Validación de la escala breve para diagnosticar estrés posttraumático (SPRINT-E) en una muestra de personas afectadas por el terremoto y tsunami del 27-F en Chile. Anales de Psicología, 29(2), 328-334.
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] Mackinnon DP, Lockwood CM, Williams J. Confidence Limits for the Indirect Effect: Distribution of the Product and Resampling Methods. Multivariate Behav Res. 2004 Jan 1;39(1):99. doi: 10.1207/s15327906mbr3901_4. PMID 20157642
- [Background] Meichenbaum, D. (1975). Self-instructional methods. En F.H. Kanfer & A.P. Goldstein (Eds.), Helping people change (pp. 357-391). New York: Pergamon Press.
- [Background] Morán C., Landero R., & González M. (2010). COPE-28: Un análisis psicométrico de la versión en español del Brief COPE. Universitas Psychologica, 9(2), 543-552.
- [Background] Morris BA, Shakespeare-Finch J. Rumination, post-traumatic growth, and distress: structural equation modelling with cancer survivors. Psychooncology. 2011 Nov;20(11):1176-83. doi: 10.1002/pon.1827. Epub 2010 Aug 23. PMID 20731009
- [Background] Moyano, E., & Ramos, N. (2007). Bienestar subjetivo: Midiendo satisfacción vital, felicidad y salud en la población chilena de la Región del Maule. Universum, 22(2), 177-193.
- [Background] Norris FH, Hamblen JL, Brown LM, Schinka JA. Validation of the Short Posttraumatic Stress Disorder Rating Interview (expanded version, Sprint-E) as a measure of postdisaster distress and treatment need. Am J Disaster Med. 2008 Jul-Aug;3(4):201-12. PMID 18822839
- [Background] Organización Mundial de la Salud (2004). Prevención de los Trastornos Mentales: Intervenciones efectivas y opciones de políticas informe compendiado. Recuperado el 20 de mayo, 2017, http://www.who.int/mental_health/evidence/Prevention_of_mental_disorders_spanish_version.pdf
- [Background] Pargament, K., Feuille, M., & Burdzy, D. (2011). The Brief RCOPE: Current psychometric status of a short measure of religious coping. Religions, 2, 51-76.
- [Background] Powers MB, Halpern JM, Ferenschak MP, Gillihan SJ, Foa EB. A meta-analytic review of prolonged exposure for posttraumatic stress disorder. Clin Psychol Rev. 2010 Aug;30(6):635-41. doi: 10.1016/j.cpr.2010.04.007. Epub 2010 May 2. PMID 20546985
- [Background] Radloff, L. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1(3), 385-401.
- [Background] Rajandram RK, Jenewein J, McGrath C, Zwahlen RA. Coping processes relevant to posttraumatic growth: an evidence-based review. Support Care Cancer. 2011 May;19(5):583-9. doi: 10.1007/s00520-011-1105-0. Epub 2011 Feb 6. PMID 21298449
- [Background] Rivera, A., & Montero, L. (2005). Espiritualidad y religiosidad en adultos mayores mexicanos. Salud Mental, 28, 51-58
- [Background] Rodríguez-Carvajal, R., Moreno-Jiménez, B. & Garrosa, E. (2006). Cuestionario de Regulación Emocional - Versión española. Madrid: Universidad Autónoma de Madrid
- [Background] Salsman JM, Segerstrom SC, Brechting EH, Carlson CR, Andrykowski MA. Posttraumatic growth and PTSD symptomatology among colorectal cancer survivors: a 3-month longitudinal examination of cognitive processing. Psychooncology. 2009 Jan;18(1):30-41. doi: 10.1002/pon.1367. PMID 18481837
- [Background] Sans-Corrales M, Pujol-Ribera E, Gene-Badia J, Pasarin-Rua MI, Iglesias-Perez B, Casajuana-Brunet J. Family medicine attributes related to satisfaction, health and costs. Fam Pract. 2006 Jun;23(3):308-16. doi: 10.1093/fampra/cmi112. Epub 2006 Feb 3. PMID 16461452
- [Background] Siqveland J, Nygaard E, Hussain A, Tedeschi RG, Heir T. Posttraumatic growth, depression and posttraumatic stress in relation to quality of life in tsunami survivors: a longitudinal study. Health Qual Life Outcomes. 2015 Feb 7;13:18. doi: 10.1186/s12955-014-0202-4. PMID 25889940
- [Background] Sutin AR, Costa PT Jr, Wethington E, Eaton W. Perceptions of stressful life events as turning points are associated with self-rated health and psychological distress. Anxiety Stress Coping. 2010 Oct;23(5):479-92. doi: 10.1080/10615800903552015. PMID 20099168
- [Background] Tedeschi RG, Calhoun LG. The Posttraumatic Growth Inventory: measuring the positive legacy of trauma. J Trauma Stress. 1996 Jul;9(3):455-71. doi: 10.1007/BF02103658. PMID 8827649
- [Background] Treynor, W., Gonzalez, R., & Nolen-Hoeksema, S. (2003). Rumination reconsidered: A psychometric analysis. Cognitive Therapy and Research, 27, 247-259.
- [Background] Vázquez, C. (2003). Técnicas cognitivas de intervención clínica. Madrid: Síntesios.
- [Background] Vazquez C, Blanco I, Sanchez A, McNally RJ. Attentional bias modification in depression through gaze contingencies and regulatory control using a new eye-tracking intervention paradigm: study protocol for a placebo-controlled trial. BMC Psychiatry. 2016 Dec 8;16(1):439. doi: 10.1186/s12888-016-1150-9. PMID 27931196
- [Background] Vázquez, C., Castilla, C. & Hervás, G. (2009). Reacciones ante el trauma: Resistencia y crecimiento. En E. Fernández-Abascal (Ed.), Las Emociones Positivas (pp. 375-392). Madrid: Pirámide.
- [Background] Wilson GT, Davison GC. Processes of fear reduction in systematic desensitization: animal studies. Psychol Bull. 1971 Jul;76(1):1-14. doi: 10.1037/h0031480. No abstract available. PMID 5105019
- [Background] Wlodarczyk, A., Basabe, N., Páez, D., Amutio, A., García, F. E., Reyes, C., & Villagrán, L. (2016). Positive effects of communal coping in the aftermath of a collective trauma: The case of the 2010 Chilean earthquake. European Journal of Education and Psychology, 9(1), 9-19.
- [Background] Wlodarczyk, A., Basabe, N., Páez, D., Villagrán, L., & Reyes, C. (2017). Individual and Collective Posttraumatic Growth in Victims of Natural Disasters: A Multidimensional Perspective. Journal of Loss and Trauma, 1-14.
- [Background] Xu J, Song X. Posttraumatic stress disorder among survivors of the Wenchuan earthquake 1 year after: prevalence and risk factors. Compr Psychiatry. 2011 Jul-Aug;52(4):431-7. doi: 10.1016/j.comppsych.2010.08.002. Epub 2010 Sep 23. PMID 21683180
- [Background] Zhou X, Wu X, Zhen R. Understanding the relationship between social support and posttraumatic stress disorder/posttraumatic growth among adolescents after Ya'an earthquake: The role of emotion regulation. Psychol Trauma. 2017 Mar;9(2):214-221. doi: 10.1037/tra0000213. Epub 2016 Oct 13. PMID 27736141
- [Background] Zoellner T, Maercker A. Posttraumatic growth in clinical psychology - a critical review and introduction of a two component model. Clin Psychol Rev. 2006 Sep;26(5):626-53. doi: 10.1016/j.cpr.2006.01.008. Epub 2006 Mar 3. PMID 16515831
- [Background] Cerna C, Garcia FE, Tellez A. Brief mindfulness, mental health, and cognitive processes: A randomized controlled trial. Psych J. 2020 Jun;9(3):359-369. doi: 10.1002/pchj.325. Epub 2019 Dec 5. PMID 31805614